CLINICAL TRIAL: NCT02880592
Title: A Multi-center, Randomized Controlled Clinical Trial Evaluating the Effect of Fresh Amniotic Membrane in the Treatment of Diabetic Foot Ulcers
Brief Title: Effect of Fresh Amniotic Membrane in the Treatment of Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Organogenesis (Industry)
Collaborators: SerenaGroup, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NT-DFU-AFF-01
Record Dates: First submitted 2016-08-23; First posted 2016-08-26 (Estimated); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Diabetic Foot Ulcers
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fresh amniotic membrane/standard of care (Experimental): This group will receive the Affinity Allograft and standard of care.
  Interventions: Other: Affinity Allograft; Other: Standard of care
- Standard of Care (Active Comparator): This group will receive standard of care for diabetic foot ulcers that includes offloading of the diabetic foot ulcer, debridement, and infection management using the appropriate dressings.
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Affinity Allograft — fresh hypothermically stored human amniotic membrane
  Arms: Fresh amniotic membrane/standard of care
Other: Standard of care — offloading, debridement, infection management using appropriate dressings

SUMMARY:
This is a multi-center, randomized controlled trial designed to evaluate the use of fresh hypothermically stored human amniotic membrane (Affinity; fHSAM) to determine if addition of fHSAM to standard of care (SOC) results in faster healing of Wagner grade 1 and 2 DFUs compared to SOC alone.

DETAILED DESCRIPTION:
This study is a multi-center, randomized, controlled open-label study designed to evaluate the safety and effectiveness of Affinity fresh amniotic membrane plus standard of care therapy (SOC) versus SOC in the treatment of diabetic foot ulcers.

The standard of care therapy in this study is offloading of the DFU, appropriate sharp or surgical debridement, and aggressive infection management. A number of offloading systems are commercially available. The choice of offloading will be at the discretion of the Principal Investigator but should be total contact casting, fixed ankle walker boot, or equivalent device to the fixed ankle walker boot.

The study will have two phases: Screening and Treatment.

The Screening Phase (1 -14 days) is designed to determine whether subjects are eligible to proceed to the Treatment Phase of the study and consists of a series of screening assessments designed to determine eligibility. At the first Screening Phase Visit, the Investigator will select the study (target) ulcer. Each subject will have only one DFU selected as the study (target) ulcer. In the situation in which a subject has more than one DFU at the S1 visit, the Investigator will select the largest DFU that meets the eligibility criteria of the protocol as the study (target) ulcer. Subjects whose target ulcer has been treated with SOC for 2 weeks are eligible to enter the treatment phase immediately once all of the inclusion and exclusion criteria are met. If the ulcer has not received SOC, the subject should be placed into SOC and enrolled in the study after 14 days of offloading.

The Treatment Phase (12 weeks) begins with a series of assessments designed to confirm the subjects' continued eligibility. Investigators will debride the ulcer, if required. Subjects whose ulcers continue to meet eligibility criteria will then be randomized to 1 of 2 groups: (1) standard of care plus weekly application of fHSAM for up to 4 weeks and thereafter per treatment guidelines (2) standard of care. During the Treatment Phase, subjects will be evaluated on a weekly basis. Efficacy evaluations each week will include Investigator assessment of ulcer healing and measurements of ulcer size using digital photos. Safety evaluations during the Treatment Phase will consist of adverse event assessments at each visit. Subject will be seen weekly (± 3 days) until the ulcer is healed or study exit if the study ulcer area has not been reduced by at least 40% within 6 weeks, or 1 week after last application treatment week 12.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old.
2. Presence of a diabetic foot ulcer, Wagner 1 or 2 grade , extending at least through the dermis or subcutaneous tissue and may involve the tendon or muscle, on any aspect of the foot provided it is below the medial aspect of the malleolus.
3. The index ulcer will be the largest ulcer if 2 or more DFUs are present with the same Wagner grade and will be the only one in the study. If other ulcerations are present on the same foot they have to be more than 2 cm apart from the index ulcer.
4. Index ulcer (i.e. current episode of ulceration) has been present for greater than 4 weeks prior to the initial screening visit and less than 1 year.
5. Study ulcer is a minimum of 0.75 cm2 and a maximum of 25 cm2 at first treatment visit.
6. Adequate circulation to the affected foot as demonstrated by a dorsum transcutaneous oxygen measurement (TCOM) or a skin perfusion pressure (SPP) measurement of ≥ 30 mmHg, or an ABI between 0.7 and 1.3 within 3 months of the first Screening Visit,or TBI of > 6 within 3 months of the first Screening Visit .
7. The target ulcer has been offloaded for at least 14 days prior to randomization.
8. Females of childbearing potential must be willing to use acceptable methods of contraception (birth control pills, barriers, or abstinence).
9. Subject understands and is willing to participate in the clinical study and can comply with weekly visits and the follow-up regimen.

Exclusion Criteria:

1. Study ulcer(s) deemed by the investigator to be caused by a medical condition other than diabetes.
2. Index ulcer, in the opinion of the investigator, is suspicious for cancer and should undergo an ulcer biopsy to rule out a carcinoma of the ulcer.
3. Subjects with a history of more than two weeks treatment with immunosuppressants (including systemic corticosteroids >10 mg daily), cytotoxic chemotherapy, or application of topical steroids to the ulcer surface within one month prior to first Screening Visit, or who receive such medications during the screening period, or who are anticipated to require such medications during the course of the study.
4. Subjects on any investigational drug(s) or therapeutic device(s) within 30 days preceding the first Screening Visit.
5. History of radiation at the ulcer site.
6. Index ulcer has been previously treated with tissue engineered materials (e.g. Apligraf® or Dermagraft®) or other scaffold materials (e.g. Oasis, Matristem) within the last 30 days preceding the first Screening Visit or will need to be treated with any prohibited therapies.
7. Affected extremity requiring negative pressure wound therapy or subject requiring hyperbaric oxygen during the course of the trial.
8. Presence of any condition(s) which seriously compromises the subject's ability to complete this study, or has a known history of poor adherence with medical treatment.
9. Osteomyelitis or bone infection of the affected foot as verified by X-ray within 30 days prior to Randomization.
10. Subject is pregnant or breast feeding.
11. Presence of diabetes with poor metabolic control as documented with an HgA1c > 12.0 within last 90 days.
12. Patients with end stage renal disease.
13. Index ulcer has reduced in area by 20% or more after 14 days of standard of care from the first screening visit (S1) to the TV1/randomization visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2016-08; Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Time to initial closure of diabetic foot ulcer | 12 weeks
  Time to initial closure of diabetic foot ulcers will be compared between the two groups.

SECONDARY OUTCOMES:
Proportion of healed wounds | 12 weeks
  The proportion of healed wounds at 12 weeks comparing the two groups.
Proportion of healed wounds | 4 weeks
  The proportion of healed wounds at 4 weeks comparing the two groups.
Quality of Life measurement | baseline and 12 weeks
  Subjects will complete the W-QoL questionnaire at baseline and 12 weeks. Changes in scores will be compared between the two groups.
Incidence of adverse events | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Katie Mowry, PhD, Study Director — NuTech Medical, Inc
Locations (8):
- United States (8):
  - GF Professional Research, Miami Lakes, Florida
  - Barry University Clinical Research, North Miami Beach, Florida
  - Henry Ford Macomb Hospital, Clinton Township, Michigan
  - Summit Health Hospital, Chambersburg, Pennsylvania
  - The Foot and Ankle Wellness Center, Ford City, Pennsylvania
  - Armstrong County Memorial Hospital, Kittanning, Pennsylvania
  - SerenaGroup Research Institute, Pittsburgh, Pennsylvania
  - Martin Foot and Ankle, York, Pennsylvania

IPD SHARING:
Plan to Share IPD: No